CLINICAL TRIAL: NCT06746246
Title: Prospective Evaluation of Multicenter Implementation of Remote Monitoring of Liver Cirrhosis Patients
Brief Title: Evaluation of Remote Monitoring of Liver Cirrhosis Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Gelre Hospitals (Other); Noordwest Ziekenhuisgroep (Other); Jeroen Bosch Ziekenhuis (Other); Albert Schweitzer Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-0284
Record Dates: First submitted 2024-12-05; First posted 2024-12-24 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2024-12

CONDITIONS: Liver Cirrhosis
Keywords: Digital health; Remote monitoring; eHealth; mHealth; Telehealth
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- 1. Standard care with remote monitoring: Liver cirrhosis patients participating in remote monitoring as part of new standard care pathway. They will give digital consent after subscription to the remote monitoring platform. Retrospective and prospective data will be gathered. Follow-up lasts 15 years, or until death.
  Patients participating in remote monitoring can be approached to give feedback about remote monitoring in terms of satisfaction, usability, applicability, compliance and feasibility.
- Standard care without remote monitoring: Liver cirrhosis patients not participating in remote monitoring. They will not be approached for informed consent and give implicit consent for data gathering unless otherwise stated in their individual electronic patient record. Retrospective and prospective data will be gathered. Follow-up lasts 15 years, or until death.

SUMMARY:
The goal of this longitudinal prospective study is to investigate disease course in patients with liver cirrhosis treated in hospitals that implemented a remote monitoring care pathway as part of their standard liver cirrhosis care pathway.

Participants will be asked to share their medical data and remote monitoring data. Therefore, this study does not contain an intervention.

ELIGIBILITY:
Inclusion Criteria:

* Liver cirrhosis diagnosis, based on liver biopsy, fibroscan (elastography), radiographic imaging and/or clinical criteria according to applied guidelines at the time of inclusion
* Age 18 years or older
* Treated at Gastroenterology department

Exclusion Criteria:

* Patients who have declined participation in scientific studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of 18 years and older with a liver cirrhosis diagnosis, treated at a Gastroenterology department in one of the participating centers.
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2040-02 (Estimated); Study Completion 2042-02 (Estimated)

PRIMARY OUTCOMES:
Number of liver related complications | From enrollment to the end of follow-up at 15 years, or untill death.
  Complications defined as: ascites, spontaneous bacterial peritonitis, variceal hemorrhage, hepatorenal syndrome, hepatopulmonary syndrome, hepatocellular carcinoma, liver failure, hepatic encephalopathy.

SECONDARY OUTCOMES:
Number of liver related clinical admissions | From enrollment to the end of follow-up at 15 years, or untill death.
  Liver related clinical admissions defined as complications related to: ascites, spontaneous bacterial peritonitis, variceal hemorrhage, hepatorenal syndrome, hepatopulmonary syndrome, hepatocellular carcinoma, liver failure, hepatic encephalopathy.
Number of liver related emergency consultations | From enrollment to the end of follow-up at 15 years, or untill death.
  Liver related emergency consultations defined as consultations due to: ascites, spontaneous bacterial peritonitis, variceal hemorrhage, hepatorenal syndrome, hepatopulmonary syndrome, hepatocellular carcinoma, liver failure, hepatic encephalopathy.
Liver transplantation | From enrollment to the end of follow-up at 15 years, or untill death.
Mortality | From enrollment to the end of follow-up at 15 years.
Number of outpatient department consultations | From enrollment to the end of follow-up at 15 years, or untill death.
  Physical or telephone
Number of liver related laboratory tests | From enrollment to the end of follow-up at 15 years, or untill death.
Number of liver related radiographic images | From enrollment to the end of follow-up at 15 years, or untill death.
Number of liver related biopsies | From enrollment to the end of follow-up at 15 years, or untill death.
Percentage of completed modules in remote monitoring sessions | From enrollment to the end of follow-up at 15 years, or untill death.

OTHER OUTCOMES:
5-level EuroQol-5 Dimensions scores | From enrollment to the end of follow-up at 15 years, or untill death.
  5-level EQ-5D version (EQ-5D-5L). The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS can be used as a quantitative measure of health outcome that reflects the patient's own judgement.

CONTACTS AND LOCATIONS:
Overall Officials: Tom Gevers, MD, PhD, Principal Investigator — Maastricht University Medical Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ganapathy D, Acharya C, Lachar J, Patidar K, Sterling RK, White MB, Ignudo C, Bommidi S, DeSoto J, Thacker LR, Matherly S, Shaw J, Siddiqui MS, Puri P, Sanyal AJ, Luketic V, Lee H, Stravitz RT, Bajaj JS. The patient buddy app can potentially prevent hepatic encephalopathy-related readmissions. Liver Int. 2017 Dec;37(12):1843-1851. doi: 10.1111/liv.13494. Epub 2017 Jul 5. PMID 28618192
- [Background] Kazankov K, Novelli S, Chatterjee DA, Phillips A, Balaji A, Raja M, Foster G, Tripathi D, Boddu R, Kumar R, Jalan R, Mookerjee RP. Evaluation of CirrhoCare(R) - a digital health solution for home management of individuals with cirrhosis. J Hepatol. 2023 Jan;78(1):123-132. doi: 10.1016/j.jhep.2022.08.034. Epub 2022 Sep 8. PMID 36087864
- [Background] de Jong MJ, van der Meulen-de Jong AE, Romberg-Camps MJ, Becx MC, Maljaars JP, Cilissen M, van Bodegraven AA, Mahmmod N, Markus T, Hameeteman WM, Dijkstra G, Masclee AA, Boonen A, Winkens B, van Tubergen A, Jonkers DM, Pierik MJ. Telemedicine for management of inflammatory bowel disease (myIBDcoach): a pragmatic, multicentre, randomised controlled trial. Lancet. 2017 Sep 2;390(10098):959-968. doi: 10.1016/S0140-6736(17)31327-2. Epub 2017 Jul 14. PMID 28716313
- [Background] Karlsen TH, Sheron N, Zelber-Sagi S, Carrieri P, Dusheiko G, Bugianesi E, Pryke R, Hutchinson SJ, Sangro B, Martin NK, Cecchini M, Dirac MA, Belloni A, Serra-Burriel M, Ponsioen CY, Sheena B, Lerouge A, Devaux M, Scott N, Hellard M, Verkade HJ, Sturm E, Marchesini G, Yki-Jarvinen H, Byrne CD, Targher G, Tur-Sinai A, Barrett D, Ninburg M, Reic T, Taylor A, Rhodes T, Treloar C, Petersen C, Schramm C, Flisiak R, Simonova MY, Pares A, Johnson P, Cucchetti A, Graupera I, Lionis C, Pose E, Fabrellas N, Ma AT, Mendive JM, Mazzaferro V, Rutter H, Cortez-Pinto H, Kelly D, Burton R, Lazarus JV, Gines P, Buti M, Newsome PN, Burra P, Manns MP. The EASL-Lancet Liver Commission: protecting the next generation of Europeans against liver disease complications and premature mortality. Lancet. 2022 Jan 1;399(10319):61-116. doi: 10.1016/S0140-6736(21)01701-3. Epub 2021 Dec 2. No abstract available. PMID 34863359
- See also: Foundation for collaborative development of e-Health tools for different chronic diseases. — https://stichtingmijncoach.nl/